CLINICAL TRIAL: NCT06776692
Title: Characterisation of Dengue Vaccine (Qdenga®, TAK-003)-Induced Humoral and Cellular Specific Immunity in Vaccinees With and Without Prior Exposure to Flavivirus Infections or Vaccination
Brief Title: Characterisation of Dengue Vaccine-induced Specific Immunity in Vaccinees With and Without Prior Exposure to Flavivirus Infections or Vaccination
Acronym: VaQDENV
Status: Recruiting | Type: Observational
Sponsor: IRCCS Sacro Cuore Don Calabria di Negrar (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-L
Record Dates: First submitted 2025-01-03; First posted 2025-01-15 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Dengue Vaccines
Keywords: Dengue; Vaccine
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: All pediatric and adult subjects attending the travel clinic of the DITM for the administration of Dengue vaccine.
  Interventions: Drug: Qdenga

INTERVENTIONS:
Drug: Qdenga — Administration of Dengue vaccine and blood sample collection

SUMMARY:
The goal of this observational study is to learn about the immunity induced by the Qdenga® vaccine in vaccinees.

Participants that will receive the Dengue vaccine as part of their routine before a travel will be asked to undergo a blood sample at the time of administration of the first dose (T0), 24-48 hours after the first dose (T1) of the vaccine, immediately before the second dose (T2 ) and one to two months after the second dose (T3). Possibly a further sample will be collected within 2 years.

DETAILED DESCRIPTION:
This is a non-profit, single-center, drug-based observational study whose primary objective is to characterize dengue-specific humoral and cellular immunity induced by the Qdenga® vaccine in vaccinees.

The study involves the enrollment of all pediatric subjects (age ≥ 4 years) and adults who present themselves at the DITM travel clinic for the administration of the Dengue vaccine; 402 patients are expected to be enrolled and will be asked to undergo a blood sample at the time of administration of the first dose (T0), 24-48 hours after the first dose (T1) of the vaccine, immediately before the second dose (T2 ) and one to two months after the second dose (T3). Possibly a further sample will be collected within 2 years (T4). The samples thus collected will be analyzed for the characterization of innate immunity, the characterization of cellular immunity and the characterization of the humoral response.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes presenting to the DITM to receive the anti-DENV vaccine whether or not they have had a history of prior DENV or other flaviviruses infection or a history of prior vaccination against other flaviviruses. These data will be recorded in the study CRF.
* Age >= 4 years.
* Signed informed consent.

Exclusion Criteria:

* Age < 4 years.
* Absence of signed informed consent.

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All pediatric and adult subjects attending the travel clinic of the DITM for the administration of Dengue vaccine will be considered eligible.
Sampling Method: Non-Probability Sample
Enrollment: 402 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Anti-DENV antibodies | BEFORE administration of the first dose (Time 0 = T0), immediately BEFORE the second dose (Time 2 = T2) of vaccine, and one to two months after the second dose (Time 3 = T3)
  Anti-DENV antibodies quantities (IgG and IgM, continuous variables unity of measure: Antibody titre dilution) BEFORE administration of the first dose (T0), immediately BEFORE the second dose (T2) of vaccine, and one to two months after the second dose (T3)

SECONDARY OUTCOMES:
Innate immunity response | BEFORE administration of the first dose (T0), after 24-48h after the first dose (Time 1 = T1)
  Type I and II IFN and IFN-inducible genes, specific cytokines and chemokines induced by Qdenga® vaccine (continuous variables: deltaCt mRNA expression and Optical Density (OD)) at T0 and T1
Cellular response | At the moment of the administration of the first dose (T0), immediately before the second dose (T2), and one to two months after the second dose (T3)
  1. immunophenotype asset: results of the flow cytometry profiles (proportions of cells),
  2. specific T- and B-cells response to viral peptides: analysis results of T- and B-cells stimulation with DENV specific peptides (continuous variables, unity of measure: Optical Density (OD)) at T0, T2 and T3.
Quantitative and qualitative anti-DENV antibody response | At the moment of the administration of the first dose (T0), immediately before the second dose (T2), and one to two months after the second dose (T3)
  1. anti-DENV antibodies quantities (IgG and IgM, continuous variables unity of measure: Antibody titre dilution) at T0, T2 and T3,
  2. Analysis results of neutralization assays against different DENV serotypes (continuous variables, unity of measure: TCID50/ml) at T0, T2 and T3,
Humoral response | At the moment of the administration of the first dose (T0), immediately before the second dose (T2), and one to two months after the second dose (T3)
  1. Analysis results humoral response against different flaviviruses (IgG and IgM, continuous variables unity of measure: Antibody titre dilution) at T0, T2 and T3,
  2. Analysis results of DENV specific avidity assays (unity of measure: Index);
  3. Previous infections with (y/n) or vaccinations against (y/n) other flaviviruses
Cell mediated response | At the moment of the administration of the first dose (T0), immediately before the second dose (T2), and one to two months after the second dose (T3)
  Analysis results cell mediated response against different flaviviruses (continuous variables, unity of measure: Optical Density (OD)) at T0, T2 and T3.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Sacro Cuore Don Calabria, Negrar, VR, Italy